CLINICAL TRIAL: NCT03964389
Title: The Effects of a Single Session of Pain Neuroscience Education (PNE) on Pain and Psychological Factors in Patients With Chronic Low Back Pain. A Double-blind Randomized Clinical Trial
Brief Title: Effectiveness of a Psychoeducative Intervention on Patients With Cronic Low Back Pain
Acronym: PNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Hospital Universitario San Juan de Alicante (Other)
Responsible Party: Principal Investigator, María Isabel Tomás Rodríguez, Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19/ 317
Record Dates: First submitted 2019-05-13; First posted 2019-05-28 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Central Nervous System Sensitization; kinesiophobia
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Intervention Model Description: two-armed randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants receive TEN sessions, but do not know that one of the groups will receive extra information
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervetion group (Experimental): A sessions of "Pain Neuroscience Education (PNE)" joint a physical exercises programs
  Interventions: Other: Pain Neuroscience Education" (PNE)
- Control group (No Intervention): Only a therapeutic physical exercises programs

INTERVENTIONS:
Other: Pain Neuroscience Education" (PNE) — A lecture on neuroscience education (EN). The aim of this intervention is to provide participants with information in a clear and simple way so that patients can change their attitude to pain, inviting them to take a more active and less contemplative role. Neuroscience has shown that it is possible to have persistent pain without tissue damage or with damage that justifies the perceived disproportion of pain.
  Other Names: Therapeutic Neuroscience Education (TNE)
  Arms: Intervetion group

SUMMARY:
One of the treatment modalities currently available in this hospital to treat this type of patients with low back pain who present with chronic pain are the group sessions that are carried out to provide information to the patient about the anatomy, biomechanics and ergonomics and are complemented with sessions of physical exercise. Based on the latest publications on treatment of this type of patients, The investigators have seen that this intervention is insufficient, and that it could be improved by combining education based on Pain Neuroscience Education (PNE)).

The present study proposes implementing this program to a randomly assigned group of patients participating in the group sessions aimed at patients with lumbar pain called "Back-pain Protocol" that are currently relized in the Physiotherapy Area of a hospital; and compare the results of this intervention with those obtained in another group that will only carry out the sessions with the traditional method that is currently used.

DETAILED DESCRIPTION:
Procedure The physiotherapist in charge of the chronic back pain programme group ("back pain protocol") is contacted. The study will be explained and the materials and training to deliver the PNE session will be provided.

Participants who meet the inclusion criteria will then be identified and randomised to the intervention or control group.

At the end of the first session, which currently takes place in group chronic back pain treatment programmes, the physiotherapist will explain the study and ask for cooperation. The information sheet is handed out. Those who decide to participate will receive an informed consent form and some questionnaires to fill in: the Numeric Pain Rating Scale (NPRS) to assess their level of pain, the Central Sensitisation Inventory, the Pain Catastrophic Scale (Spanish version), the Tampa Kinesiofobia Scale (TSK).

Interventions The current protocol consists of five sessions spread over one and a half months. Patients come to the rehabilitation classroom in two groups of 10 people per day for one hour.

The first session consists of an informative talk. The physiotherapist gives information and explanations about the "back pain protocol". The physiotherapist explains the problems of posture and gestures that can be beneficial or detrimental to their treatment, their daily activities, their work and their sporting activities.

In the second, third and fourth sessions, the participants learn specific exercises for back pain. Patients receive a booklet with the exercises and postures to be incorporated into their daily habits.

Treatment. This study proposes that only participants assigned to the intervention group will also receive an additional patient education session on Pain Neuroscience Education (PNE).

This session will last one hour and will be given in an additional session the day after the first information session of the current protocol. They will also be given information to read and review at home. Only patients randomised to the intervention group will attend this session.

The aim of this intervention is to provide participants with information in a clear and simple way, so that they can change their attitude to pain, inviting them to take a more active and less contemplative role. The physiotherapist will explain to the participants in a simple way that chronic pain is not always the result of tissue damage. Neuroscience has shown that it is possible to have persistent pain without tissue damage or with damage that justifies the perception of disproportionate pain. The physiotherapist will also explain the difference between acute and chronic pain, central sensitisation processes (CS) and endogenous pain control mechanisms. The physiotherapist will talk about how thoughts, beliefs and emotions modify the painful experience and how the erroneous information received, sometimes iatrogenic, modifies the mechanisms of pain processing. The content of the neuroscience education lectures is based on the book Explain Pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in the "back protocol" groups in the hospital
* That present pain of more than 3 months of evolution

Exclusion Criteria:

* Oncological pain
* Fracture or spinal surgery in the last year
* Cognitive neurological alteration that prevents understanding the contents of the session
* Alterations at the motor level that prevent the realization of the program of directed physical exercise that is currently carried out
* Pregnancy
* Urinary or intestinal incontinence
* Other clinical conditions that may aggravate chronic spinal pain (chronic fatigue syndrome, fibromyalgia and complex regional pain syndrome)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 weeks following the reported onset of symptoms.
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")

SECONDARY OUTCOMES:
Pain Catastrophizing: Pain Catastrophizing Scale | baseline, 5 weeks and 12 weeks
  Pain Catastrophizing Scale. Catastrophic thinking has widely been recognized in the development and maintenance of hypochondriasis and anxiety disorders.The PCS is a 13 item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). The PCS is broken into three subscales being magnification, rumination, and helplessness. The scale was developed as a self-report measurement tool that provided a valid index of catastrophizing in clinical and non-clinical populations. ranges from '0' representing no pain catastrophizing to '52' representing maximum pain catastrophizing
Kinesiophobia: Tampa Scale for Kinesiophobia (TSK 11) | baseline, 5 weeks and 12 weeks
  Tampa Scale of Kinesiophobia (TSK-11) . It assesses the fear of a patient related with suffering a re-injury again during movement through 11 items. With a score range of 11 to 44, the TSK-11 has demonstrated acceptable internal consistency and validity. A 4-point reduction optimally identifies an significant reduction in the fear of the patient associated with the movement and presents a minimal detectable change of 5.60 points
- Central sensitisation inventory (CSI) | baseline, 5 weeks and 12 weeks
  This instrument is proposed to identify a potential CS syndrome in patients and to assess comorbidities associated with chronic pain, according to the IASP criterio. It contains 25 items scored on a Likert-type scale from 0 to 4. Total score ranges from 0 to 100, with a set cut-off of 40 points to differentiate subjects with and without potential CS or to confirm the presence of pain comorbidities (sensitivity: 85%, specificity: 75%) [32]. Recently, severity ranges have been proposed for CS: subclinical (0-29), mild (30-39), moderate (40-49), severe (50-59) and extreme (60-100).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de San Juande Alicante, Sant Joan d'Alacant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Traeger AC, Lee H, Hubscher M, Skinner IW, Moseley GL, Nicholas MK, Henschke N, Refshauge KM, Blyth FM, Main CJ, Hush JM, Lo S, McAuley JH. Effect of Intensive Patient Education vs Placebo Patient Education on Outcomes in Patients With Acute Low Back Pain: A Randomized Clinical Trial. JAMA Neurol. 2019 Feb 1;76(2):161-169. doi: 10.1001/jamaneurol.2018.3376. PMID 30398542
- See also: Learn a science based approach to overcome chronic pain. — https://www.retrainpain.org/
- See also: An international research group that focuses on pain an dody movement — http://www.paininmotion.be/